CLINICAL TRIAL: NCT03731819
Title: Establishment of Abbreviated Pancreatobiliary MRI Using Compressed Sensing Technique for Pancreas Cystic Neoplasm Follow-up
Brief Title: Establishment of Abbreviated Pancreatobiliary MRI Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Hee Yoon, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNUH-2018-1276
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Pancreas Cyst; Intraductal Papillary Mucinous Neoplasm
Keywords: MRI
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follow-up participants (Experimental): Patients who met eligibility criteria. Participants are going to undergo Abbreviated PB MRI.
  Interventions: Diagnostic Test: Abbreviated PB MRI

INTERVENTIONS:
Diagnostic Test: Abbreviated PB MRI — Abbreviated PB MRI which targets table time of 10 minutes. For MRI acquisition, standard dose of commercially available MR contrast agent (Gadovist, Bayer, Germany) is used on weight-based dosing (0.1mmol/kg).

SUMMARY:
This study aims to establish abbreviated PB MRI protocol for patients on regular imaging follow-up for pancreas cystic neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* on follow-up for pancreas intraductal mucinous neoplasm
* OR incidentally detected pancreas cyst (equal to or larger than 1cm)
* AND scheduled for CECT or has CECT within a months
* AND sign informed consent

Exclusion Criteria:

* Any absolute or relative contra-indication for contrast-enhanced MRI
* No pancreas cystic neoplasm
* History of pancreatectomy
* History of any procedure for pancreatic cyst (ablation, aspiration...) in a year
* Hemosiderosis
* Suspicion of acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Table time of Abbreviated PB MRI | 1 day after PB MRI acquisition
  total scan time

SECONDARY OUTCOMES:
In room time of Abbreviated PB MRI | 1 day after PB MRI acquisition
  time spent in room by participants (difference between walk-in and walk-out times)
Diagnostic confidence | 6 months after participants enrollment
  subjective diagnostic confidence for pancreas cystic neoplasm on five point scale
Image quality | 6 months after participants enrollment
  overall image quality of Abbreviated PB MRI
Requirement for re-examination | 6 months after participants enrollment
  clinical need for re-examination due to suboptimal image quality

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hee Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No